CLINICAL TRIAL: NCT06069999
Title: Bedside Telerehabilitation Early After CNS Injury
Brief Title: Telerehabilitation Early After CNS Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRCare, Inc. (Industry)
Collaborators: California Rehabilitation Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRC-09
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Stroke; Traumatic Brain Injury; Spinal Cord Injuries
Keywords: Stroke; Traumatic Brain Injuries; Spinal Cord Injuries; Telerehabilitation; Brain Plasticity; Telehealth
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TR Bedside Telerehabilitation (Experimental): Participants will be assigned 45-minutes of therapy training exercises each day for 7 days a week up to 4 weeks or until discharge.
  Participants will use the HandyMotion device to interact with the telerehabilitation program displayed on the TV set in the patient room.
  Interventions: Device: HandyMotion Treatment Program

INTERVENTIONS:
Device: HandyMotion Treatment Program — A pair of sensor-based wireless remote controllers to allow the performance of functional exercises and games that target arm movement.

SUMMARY:
The goal of this clinical trial is to assess the safety and feasibility of providing extra doses of rehabilitation therapy for persons with a recent stroke, traumatic brain injury (TBI) and/or spinal cord injury (SCI). The therapy treatment targets to improve arm function by introducing telerehabilitation to the bedside of participants during the inpatient rehab admission period. Participants will use a newly developed functional training system (HandyMotion) to access therapy treatment program directly from their hospital room. HandyMotion is a sensor-based training system that can connect to the TV set in the hospital room, enabling patients to access their therapy training program to practice rehab-oriented games and exercises ad libitum, at any time of the day.

DETAILED DESCRIPTION:
This clinical trial is designed to address 3 specific aims:

Aim 1: To measure the safety of daily bedside telerehabilitation.

Aim 2: To measure the feasibility of daily bedside telerehabilitation.

Aim 3: To derive a preliminary estimate of motor and functional outcomes in patients engaged in daily bedside telerehabilitation. This is an uncontrolled pilot study, and so it is understood that such measures cannot be attributed to the telerehabilitation intervention, however, these measures will describe the clinical course of a patient engaged in this intervention.

Telerehabilitation therapy is delivered over the course of the inpatient rehabilitation stay. A therapist-facing web portal is used for treatment planning and patient monitoring. The treatment approach was initially designed based on an upper-extremity task-specific training manual and Accelerated Skill Acquisition Program.

Each daily 45-minute treatment session is created by a licensed OT or PT and includes:

A. At least 15 min/day of upper extremity exercises. In addition, therapists have the option to incorporate standard exercise equipment (e.g., Theraband or dowels) that can be incorporated into assigned exercises.

B. At least 15 min/day of functional training through games. The study provides 2 controllers with 5 different input devices that are available to drive game play. Games stress various motor control features (e.g., varying movement speed, range of motion, target size, extent of visuomotor tracking, or level of cognitive demand), which are selected and adjusted by the therapist.

C. If applicable, 5 minutes/day of stroke education. The education content targets five categories (Stroke Risk Factors, Stroke Prevention, Effects of Stroke, Diet, and Exercise) and corresponds to the Stroke Knowledge Exam.

The remaining 10-15 minutes consist of additional exercises and games, per the judgment of the licensed OT or PT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. CNS injury with onset in the prior 90 days

   1. For stroke: Stroke that is radiologically verified and due to ischemia or to intracerebral hemorrhage.
   2. For traumatic brain injury: History that is consistent with TBI; and score on the Revised Rancho Levels of Cognitive Functioning Scale is at least 6 out of 10.
   3. For spinal cord injury: Traumatic or nontraumatic, incomplete cervical SCI.
3. At least one arm must have motor deficits that are neither very mild nor devastating (dense arm plegia). Operationally, this requires that the Visit 1 Box & Block Test score is at least 1 block, but no more than 30 blocks, in 60 seconds.
4. Possess enough arm movement to participate in therapy, including able to hold the HandyMotion device in the paretic hand(s), using an assistive device if needed.
5. Informed consent signed by the subject (no surrogate consent permitted for this study)
6. Able to follow simple instructions
7. Study participation is not likely to be significantly limited by agitated behavior

Exclusion Criteria:

1. A major, active, coexistent neurological or psychiatric disease that would limit study participation, e.g., advanced dementia or active psychosis
2. Expectation that patient's cognitive status will likely interfere substantially with playing assigned games or exercises
3. Deficits in communication that interfere with reasonable study participation
4. Lacking visual acuity, with or without corrective lens, of 20/50 or better in at least one eye
5. Subject does not speak sufficient English to comply with study procedures
6. Shoulder pain that in the judgement of the study team is likely to substantially limit the amount of TR therapy completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of daily beside telerehabilitation based on incidence of treatment-emergent adverse events as assessed by regular review of the medical record and patient interview | "For approximately 4 weeks, up until discharge"
  Safety will be measured in terms of adverse events (AEs) deemed related to use of the telerehabilitation system on a probable or definite basis.

SECONDARY OUTCOMES:
Feasibility of daily bedside telerehabilitation based on measurement of patient compliance, as determined by reviewing electronic records of device usage | "baseline" and "immediately after end of treatment"
  Feasibility will be measured in terms of patient compliance, specifically the fraction of days where a patient is assigned to do bedside telerehabilitation and initiates a treatment session. Any factors related to reduced compliance, including technical and medical factors, will be recorded.
  Feasibility is a composite measure. It is descriptive, so that all of these observations can be combined into a single outcome.
Box and Blocks Test | "baseline" and "immediately after end of treatment"
  Measure of Upper Extremity Function by assessing unilateral gross manual dexterity.
  Participants will be asked to perform the test twice for each side to assess bilateral gross manual dexterity. Participants will be asked to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Su, MD, Principal Investigator — California Rehabilitation Institute
Locations (5):
- United States (5):
  - California Rehabilitation Institute, Los Angeles, California
  - Casa Colina Hospital and Centers for Healthcare, Pomona, California
  - Brooks Rehabilitation, Jacksonville, Florida
  - Jefferson Moss-Magee Rehabilitation, Philadelphia, Pennsylvania
  - University of Utah - Craig H. Neilsen Rehabilitation Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No